CLINICAL TRIAL: NCT02646332
Title: Comparing the Efficacy and Impact on Gastrointestinal Microbiota of Reverse Hybrid Therapy and Concomitant Therapy in Helicobacter Pylori Eradication
Brief Title: Comparing the Efficacy of Reverse Hybrid Therapy and Concomitant Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS15-CT7-15
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate
MeSH Terms: interventions — Amoxicillin; Clarithromycin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (dexlan+amox+clar+metr)+(dexlan+amox) (Experimental): a 7-day quadruple regimen with dexlansoprazole MR 60 mg once daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily, followed by a 7-day dual regimen with dexlansoprazole MR 60 mg once daily and amoxicillin 1 g twice daily
  Interventions: Drug: (dexlan+amox+clar+metr)+(dexlan+amox)
- dexlan+clarith+amox+metro (Active Comparator): dexlansoprazole MR 60 mg once daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily for 14 days
  Interventions: Drug: dexlan+clarith+amox+metro

INTERVENTIONS:
Drug: (dexlan+amox+clar+metr)+(dexlan+amox) — a 7-day quadruple regimen with dexlansoprazole MR 60 mg once daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily, followed by a 7-day dual regimen with dexlansoprazole MR 60 mg once daily and amoxicillin 1 g twice daily
  Other Names: dexlansoprazole MR 60 mg; amoxicillin 1 g; clarithromycin 500 mg; metronidazole 250 mg
  Arms: (dexlan+amox+clar+metr)+(dexlan+amox)
Drug: dexlan+clarith+amox+metro — dexlansoprazole MR 60 mg once daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily for 14 days
  Other Names: dexlansoprazole MR 60 mg; clarithromycin 500 mg; amoxicillin 1 g; metronidazole 250 mg
  Arms: dexlan+clarith+amox+metro

SUMMARY:
Reverse hybrid therapy achieves a higher eradication rate than concomitant therapy remains unanswered.

DETAILED DESCRIPTION:
A 14-day hybrid therapy invented by our study group appears very promising in H. pylori eradication, achieving excellent eradication rates of 99% and 97% according to per-protocol and intention-to-treat analyses, respectively. Recently, the investigators demonstrated that the eradication rate of reverse hybrid therapy was higher than that of standard triple therapy. However, whether reverse hybrid therapy achieves a higher eradication rate than concomitant therapy remains unanswered.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2015-12; Primary Completion 2020-07-31 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | (Dexlan+Amox+Clar+Metr)+(Dexlan+Amox) | Dexlan+Clarith+Amox+Metro
Started | 124 | 124
Completed | 124 | 121
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (Dexlan+Amox+Clar+Metr)+(Dexlan+Amox) | Dexlan+Clarith+Amox+Metro | Total
Number analyzed (Participants) | 124 | 124 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.3) | 54.7 (11.2) | 55.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 64 | 130
  Male | 58 | 60 | 118
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 124 | 124 | 248
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 124 | 124 | 248
History of smoking [Number; unit: participants] | 18 | 26 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: To assess eradication efficacy,repeated endoscopy with rapid urease test, histological examination and culture or Urea breath test.
Time Frame: sixth week after the end of anti- H. pylori therapy
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | (Dexlan+Amox+Clar+Metr)+(Dexlan+Amox) | Dexlan+Clarith+Amox+Metro
Number analyzed (Participants) | 124 | 124
participants | 124 | 121

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | (Dexlan+Amox+Clar+Metr)+(Dexlan+Amox) | Dexlan+Clarith+Amox+Metro
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/124
Serious Adverse Events (participants affected / at risk) | 0/124 | 0/124
Other Adverse Events (participants affected / at risk) | 25/124 | 48/124
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (Dexlan+Amox+Clar+Metr)+(Dexlan+Amox) (N=124) | Dexlan+Clarith+Amox+Metro (N=124)
Nausea (Gastrointestinal disorders) | 11 (11) | 13 (13)
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 23 (23)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 6 (6)
Skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6)

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02646332/Prot_SAP_000.pdf